CLINICAL TRIAL: NCT01526759
Title: The Effect of 2 Weeks of Supplementation of a High-gelling, High-viscous Dietary Fibre on Energy Intake
Brief Title: Fiber Longer Term Study on Energy Intake
Acronym: FLiTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NL38515.081.11
Record Dates: First submitted 2011-12-23; First posted 2012-02-06 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: dietary fiber; energy intake; satiety; physicochemical properties; men and women; Healthy adults
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Gelatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pectin (Experimental): 10 gram high gelling-high viscous fiber, added to a drink
  Interventions: Dietary Supplement: LM pectin (10%)
- control (Placebo Comparator): 10g gelatin, added to a drink
  Interventions: Dietary Supplement: gelatin

INTERVENTIONS:
Dietary Supplement: LM pectin (10%) — 15 days 1 daily consumption of a drink with 10g pectin added
  Arms: pectin
Dietary Supplement: gelatin — 15 days 1 daily consumption of a drink with 10g gelatin added
  Arms: control

SUMMARY:
Dietary fibre seems to have a relevant role in body weight management. In an acute study the investigators found that high viscous-high gelling pectin increased feelings of satiety. The objective of this study is to study the effects of 2 weeks of supplementation of high gelling-high viscous fibre or a high gelling-high viscous non-fibre control on energy intake.

The investigators do this by measuring the difference in ad libitum energy intake after 15 days of pectin or 15 days of control supplements. The investigators will further measure differences in 24h feelings of satiety, fasting blood glucose and insulin, fermentation and composition of microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-30 year
* BMI: 18.5-25 kg/m2
* Healthy: as judged by the participant
* H2 producer

Exclusion Criteria:

* Weight loss or weight gain of more than 5 kg during the last 2 months
* Using an energy restricted diet during the last 2 months
* Lack of appetite for any reason
* Restrained eater
* Smoking
* Heavy alcohol use: >5 drinks/day
* Reported stomach or bowel diseases or disorders (e.g. irritable bowel syndrome)
* Reported diabetes
* Reported thyroid disease or any other endocrine disorder
* Using medication other than birth control, paracetamol, aspirin, hey fever and asthma
* Antibiotic use <2 months before the study
* Reported intolerance, allergy, or not liking of the research foods
* Vegetarian
* Current dietary fibre supplementation
* Fasting glucose levels >5.8 mmol/l
* Experienced any problems with drawing blood in the past
* Thesis students or employees of the division of Human Nutrition
* Volunteers who participated in the ProVe study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Energy intake | change from placebo after 2 weeks
  after 14 days of both intervention and placebo supplements ad libitum energy intake is measured for 3 days in a row. The change in energy intake will be calculated.

SECONDARY OUTCOMES:
satiety | change from placebo after 1 day and 15 days
  at day 1 and after 15 days of both supplement and placebo intake satiety is measured hourly over 1 day at waking hours. The change in satiety will be calculated.
fasting glucose | change from placebo after day 0, 1 and 15
  at day 0, 1 and day 15 of supplementation period fasting glucose is measured
fasting insulin | change from placebo after day 0, 1 and 15
  at day 0, 1 and day 15 of supplementation period fasting insulin is measured
fasting leptin | change from placebo after day 0, 1 and 15
  at day 0, 1 and day 15 of supplementation period fasting leptin is measured
hydrogen in breath | change from placebo after day 2 and 15
  at day 2 and at day 15 hydrogen is measured hourly over 1 day at waking hours
energy intake | change from placebo after day 0 and 1
  before supplement intake and after 1 day of supplement 1-day ad libitum energy intake is measured. The change in energy intake will be calculated.
body weight | change from placebo after day 0,1,2,14,15, 16 and 17
  Each day the subject reports to the research center, body weight is measured. The change in body weight compared to placebo will be calculated.
adverse events | daily from day 0 to day 16
  participants will be asked to register adverse events daily in a diary. They are also asked to report ae's to the researchers. number and type of AEs after fibre supplements will be compared to number and type of AEs after placebo supplements

CONTACTS AND LOCATIONS:
Overall Officials: Edith Feskens, Prof, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Netherlands